CLINICAL TRIAL: NCT02064244
Title: Does the Inferior Vena Cava Size Assessment Help in the Management of Acute Kidney Injury in Critically Ill Patients?
Brief Title: Inferior Vena Cava (IVC) Size in Acute Renal Failure
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 3464
Record Dates: First submitted 2014-02-06; First posted 2014-02-17 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Acute Renal Failure
Keywords: renal; kidney; creatinine; Inferior Vena Cava (IVC); Acute Renal Failure (ARF); Acute Kidney Injury (AKI)
MeSH Terms: conditions — Acute Kidney Injury | interventions — High-Energy Shock Waves

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute renal failure in ICU: Ultrasound for measurement of Inferior Vena Cava size
  Interventions: Other: Ultrasound for measurement of Inferior Vena Cava size.

INTERVENTIONS:
Other: Ultrasound for measurement of Inferior Vena Cava size. — Focused bedside ultrasound will be performed for each patient as part of their routine care and initial assessment. The IVC size will be measured at the subcostal window, during inspiration and expiration, using the Sonosite cardiac probe P-21 (5-1 MHZ). The measurement is obtained by applying the M-mode, perpendicular to the IVC axis and 2 cm caudal from its junction with the right atrium.

SUMMARY:
Bedside ultrasonographic assessment of IVC size and IVC collapsibility index can be used to guide the management of patients with acute kidney injury with and without volume overload in the intensive care unit

DETAILED DESCRIPTION:
Consecutive patients presenting to the intensive care unit with a diagnosis of acute renal failure (defined as a 1.5 fold increase in plasma Creatinine level compared to baseline ).

Baseline characteristics will be recorded and followed for each patient, these include:

1. Demographics
2. Medical history
3. Hemodynamic parameter such as Central Venous Pressure (CVP), Mean Arterial Pressure (MAP) , and measurement of superior vena cava (SVC) size by ultrasound.
4. Laboratory parameter such as chemistry, fractional excretion of sodium , fractional excretion of urea , beta natriuretic peptide , albumin
5. Radiographic parameters
6. Echocardiographic parameters including Left Ventricular Ejection Fraction (LVEF), Right Ventricular (RV) function and IVC size and variations
7. Mechanical ventilation
8. Daily fluid balance

Focused bedside ultrasound will be performed for each patient as part of their routine care and initial assessment. The IVC size will be measured at the subcostal window, during inspiration and expiration, using the (Sonosite) Cardiac probe P-21 (5-1 MHZ). The measurement is obtained by applying the M-mode, perpendicular to the IVC axis and 2 cm caudal from its junction with the right atrium.

In spontaneously breathing, non-ventilated patients, we will calculate the IVC collapsibility index (IVC-CI) = [IVC max-IVC min]/IVC max.

Whereas in patients who are mechanically ventilated we will calculate their IVC variation index (ΔIVC) = IVC max-IVC min/ IVC mean diameter.

IVC-CI, ΔIVC, IVC size will be used to classify patient as volume responders or non-responder. Prior studies have suggested Intravascular volume depletion is likely present when the, IVC<1 cm , IVC-CI is > 50% in spontaneously breathing patients and volume responsiveness when the ΔIVC is ≥ 12% in mechanically ventilated patient .

The Fractional excretion of sodium as well as the fractional excretion of urea (when diuretics are used) will be calculated to classify the etiology of the renal failure as pre-renal or intrinsic renal failure.

Fluid balance as well as the change in plasma Creatinine level at 48 hours post admission will be recorded.

Two groups of patients will be identified:

* Group 1 includes the patients who were managed in concordance with their IVC measurements (Volume responders who had a positive fluid balance at 48 h post admission and volume non responders who had an even or negative fluid balance at 48 hours post admission).
* Group 2 includes the patients in whom the fluid management was discordant with the IVC measurement.

Analyses will be done at 24 as well as 48 hours post admission.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the intensive care unit with a diagnosis of acute renal failure (defined as a 1.5 fold increase in plasma Creatinine level compared to baseline)

Exclusion Criteria:

* Age<18 years
* Hemodialysis or continuous renal replacement therapy(CRRT)
* Untreated obstructive uropathy
* Pulmonary emboli

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting to the intensive care unit with a diagnosis of acute renal failure ( Defined as 1.5 fold increase in plasma creatinine level compared to baseline)
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
percentage of patients with improved Creatinine level in group 1 and 2 | 48 hours
  percentage of patients with improved Creatinine level in group 1 and 2

SECONDARY OUTCOMES:
glomerular filtration rate (GFR), changes in hemodynamic parameters (mean arterial blood pressure, urine output, pressors requirement )and Partial oxygen pressure (PO2) /Fio2 in group 1 and group 2 | 24 and 48 hours
  glomerular filtration rate (GFR), changes in hemodynamic parameters (mean arterial blood pressure, urine output, pressors requirement) and Partial O2 /Fio2 in group 1 and group 2.
  Different cut off for IVC size measurement and variations will be used to improve the predictive value of the ultrasound in the management of renal failure in hypervolemic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Houssein Youness, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Jambeih R, Keddissi JI, Youness HA. IVC Measurements in Critically Ill Patients with Acute Renal Failure. Crit Care Res Pract. 2017;2017:3598392. doi: 10.1155/2017/3598392. Epub 2017 Sep 5. PMID 29057120